CLINICAL TRIAL: NCT06435559
Title: CHEMioterapia e Deterioramento cOgnitivo Nelle Pazienti aFfette da Carcinoma Mammario
Brief Title: CHEmotherapy and Cognitive Deterioration in Patients With Operable Breast Cancer: Impact of Cognitive Rehabilitation (CHEMOFOG)
Acronym: CHEMOFOG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHEMOFOG
Record Dates: First submitted 2024-05-19; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
Keywords: Chemotherapy-induced cognitive impairment; Neuropsychological assessments; Breast cancer; Adjuvant chemotherapy; Neo-adjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Chemotherapy-Related Cognitive Impairment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A-experimental group (Experimental): Patient enrolled in a cognitive rehabilitation program using Neurotablet® and paper and pencil exercises
  Interventions: Other: Neurotablet® and Neuropsychological evaluations
- B-control group (Other): Patient NOT enrolled in a cognitive rehabilitation program using Neurotablet® and paper and pencil exercises.
  Interventions: Other: Neuropsychological evaluations

INTERVENTIONS:
Other: Neurotablet® and Neuropsychological evaluations — The experimental group will carry out cognitive rehabilitation using the Neurotablet device. The cognitive rehabilitation will be performed for 10 consecutive weeks, once a week for 1 hour. Neuropsychological evaluations will be conducted before the start of chemotherapy (T0), 6 months (T1) and 12 months (T2) after the start of chemotherapy. Neuropsychological evaluations will include tests to analyze the main cognitive domains of memory, attention, executive functions and learning.
  Arms: A-experimental group
Other: Neuropsychological evaluations — Neuropsychological evaluations will be conducted before the start of chemotherapy (T0), 6 months (T1) and 12 months (T2) after the start of chemotherapy. Neuropsychological evaluations will include tests to analyze the main cognitive domains of memory, attention, executive functions and learning.
  Arms: B-control group

SUMMARY:
An interventional, non-pharmacological, monocentric study evaluating the effectiveness of cognitive rehabilitation in counteracting chemotherapy-induced cognitive impairment (CRCI) in women with operable breast cancer treated with neo-adjuvant therapy and/ or adjuvant therapy.

DETAILED DESCRIPTION:
This interventional, non-pharmacological, monocentric study examines the effectiveness of cognitive rehabilitation in counteracting CRCI in women with operable breast cancer treated with neo-adjuvant therapy and/ or adjuvant therapy.

A total of 128 patients will be randomized 1:1 into two groups:

* Experimental group, which will participate in a cognitive rehabilitation program using Neurotablet® and paper and pencil exercises. To evaluate the efficacy of the cognitive rehabilitation program, neurocognitive evaluations will be performed.
* Control group, which will only carry out neuropsychological assessments.

Neuropsychological evaluations will be conducted before the start of chemotherapy (T0), 6 months (T1) and 12 months (T2) after the start of chemotherapy. Neuropsychological evaluations will include tests to analyze the main cognitive domains of memory, attention, executive functions and learning.

ELIGIBILITY:
Inclusion Criteria:

* Signature of informed consent
* Diagnosis of operable/operated breast cancer
* Patients candidate to be treated with Neo/adjuvant chemotherapy

Exclusion Criteria:

* Previous chemotherapy treatments
* Patients with Metastatic breast cancer
* Patients affected by pathologies of the brain, head trauma, and intellectual disabilities
* Patients affected by previous or current neurological and/or psychiatric disorders
* Patients currently treated with psychopharmacological drug

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of a 10-week cognitive rehabilitation program | Neurocognitive evaluations will be performed at T0 (before chemotherapy program start), T1 (after 6 months from chemotherapy started), and T2 (after 12 months from chemotherapy started)
  Test the effectiveness of a 10-week cognitive rehabilitation program in limiting or preventing chemotherapy-induced cognitive impairment. To test the efficacy of this cognitive rehabilitation program, neurocognitive evaluations will be performed.

SECONDARY OUTCOMES:
Analysis of cognitive function trends in the control group | Neurocognitive evaluations will be performed at T0 (before chemotherapy program start), T1 (after 6 months from chemotherapy started), and T2 (after 12 months from chemotherapy started)
  Analysis of cognitive function trends though neurocognitive evaluations

CONTACTS AND LOCATIONS:
Overall Officials: Ornella Garrone, MD, Principal Investigator — Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico-SC Oncologia Medica

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lauby-Secretan B, Scoccianti C, Loomis D, Benbrahim-Tallaa L, Bouvard V, Bianchini F, Straif K; International Agency for Research on Cancer Handbook Working Group. Breast-cancer screening--viewpoint of the IARC Working Group. N Engl J Med. 2015 Jun 11;372(24):2353-8. doi: 10.1056/NEJMsr1504363. Epub 2015 Jun 3. No abstract available. PMID 26039523
- [Background] Rodriguez Martin B, Fernandez Rodriguez EJ, Rihuete Galve MI, Cruz Hernandez JJ. Study of Chemotherapy-Induced Cognitive Impairment in Women with Breast Cancer. Int J Environ Res Public Health. 2020 Nov 30;17(23):8896. doi: 10.3390/ijerph17238896. PMID 33265966
- [Background] Wefel JS, Saleeba AK, Buzdar AU, Meyers CA. Acute and late onset cognitive dysfunction associated with chemotherapy in women with breast cancer. Cancer. 2010 Jul 15;116(14):3348-56. doi: 10.1002/cncr.25098. PMID 20564075
- [Background] Ercoli LM, Petersen L, Hunter AM, Castellon SA, Kwan L, Kahn-Mills BA, Embree LM, Cernin PA, Leuchter AF, Ganz PA. Cognitive rehabilitation group intervention for breast cancer survivors: results of a randomized clinical trial. Psychooncology. 2015 Nov;24(11):1360-7. doi: 10.1002/pon.3769. Epub 2015 Mar 10. PMID 25759235
- [Background] Hurria A, Somlo G, Ahles T. Renaming "chemobrain". Cancer Invest. 2007 Sep;25(6):373-7. doi: 10.1080/07357900701506672. PMID 17882646
- [Background] Argyriou AA, Assimakopoulos K, Iconomou G, Giannakopoulou F, Kalofonos HP. Either called "chemobrain" or "chemofog," the long-term chemotherapy-induced cognitive decline in cancer survivors is real. J Pain Symptom Manage. 2011 Jan;41(1):126-39. doi: 10.1016/j.jpainsymman.2010.04.021. Epub 2010 Sep 15. PMID 20832978
- [Background] Sioka C, Kyritsis AP. Central and peripheral nervous system toxicity of common chemotherapeutic agents. Cancer Chemother Pharmacol. 2009 Apr;63(5):761-7. doi: 10.1007/s00280-008-0876-6. Epub 2008 Nov 25. PMID 19034447
- [Background] Vezmar S, Schusseler P, Becker A, Bode U, Jaehde U. Methotrexate-associated alterations of the folate and methyl-transfer pathway in the CSF of ALL patients with and without symptoms of neurotoxicity. Pediatr Blood Cancer. 2009 Jan;52(1):26-32. doi: 10.1002/pbc.21827. PMID 19006245
- [Background] Vardy J, Dhillon H. The fog hasn't lifted on "chemobrain" yet: ongoing uncertainty regarding the effects of chemotherapy and breast cancer on cognition. Breast Cancer Res Treat. 2010 Aug;123(1):35-7. doi: 10.1007/s10549-009-0719-0. Epub 2010 Jan 6. No abstract available. PMID 20052534
- [Background] Iconomou G, Mega V, Koutras A, Iconomou AV, Kalofonos HP. Prospective assessment of emotional distress, cognitive function, and quality of life in patients with cancer treated with chemotherapy. Cancer. 2004 Jul 15;101(2):404-11. doi: 10.1002/cncr.20385. PMID 15241840
- [Background] Hurria A, Rosen C, Hudis C, Zuckerman E, Panageas KS, Lachs MS, Witmer M, van Gorp WG, Fornier M, D'Andrea G, Moasser M, Dang C, Van Poznak C, Hurria A, Holland J. Cognitive function of older patients receiving adjuvant chemotherapy for breast cancer: a pilot prospective longitudinal study. J Am Geriatr Soc. 2006 Jun;54(6):925-31. doi: 10.1111/j.1532-5415.2006.00732.x. PMID 16776787
- [Background] Von Ah D, Crouch A. Cognitive Rehabilitation for Cognitive Dysfunction after Cancer and Cancer Treatment: Implications for Nursing Practice. Semin Oncol Nurs. 2020 Feb;36(1):150977. doi: 10.1016/j.soncn.2019.150977. Epub 2020 Jan 17. PMID 31959511
- [Background] Bray VJ, Dhillon HM, Bell ML, Kabourakis M, Fiero MH, Yip D, Boyle F, Price MA, Vardy JL. Evaluation of a Web-Based Cognitive Rehabilitation Program in Cancer Survivors Reporting Cognitive Symptoms After Chemotherapy. J Clin Oncol. 2017 Jan 10;35(2):217-225. doi: 10.1200/JCO.2016.67.8201. Epub 2016 Oct 28. PMID 28056205
- [Background] Von Ah D. Cognitive changes associated with cancer and cancer treatment: state of the science. Clin J Oncol Nurs. 2015 Feb;19(1):47-56. doi: 10.1188/15.CJON.19-01AP. PMID 25689649
- [Background] Foderaro G, Isella V, Mazzone A, Biglia E, Di Gangi M, Pasotti F, Sansotera F, Grobberio M, Raimondi V, Mapelli C, Ferri F, Impagnatiello V, Ferrarese C, Appollonio IM. Brand new norms for a good old test: Northern Italy normative study of MiniMental State Examination. Neurol Sci. 2022 May;43(5):3053-3063. doi: 10.1007/s10072-021-05845-4. Epub 2022 Jan 6. PMID 34989910
- [Background] Monaco M, Costa A, Caltagirone C, Carlesimo GA. Forward and backward span for verbal and visuo-spatial data: standardization and normative data from an Italian adult population. Neurol Sci. 2013 May;34(5):749-54. doi: 10.1007/s10072-012-1130-x. Epub 2012 Jun 12. PMID 22689311
- [Background] Conca F, Esposito V, Rundo F, Quaranta D, Muscio C, Manenti R, Caruso G, Lucca U, Galbussera AA, Di Tella S, Baglio F, L'Abbate F, Canu E, Catania V, Filippi M, Mattavelli G, Poletti B, Silani V, Lodi R, De Matteis M, Stanzani Maserati M, Arighi A, Rotondo E, Tanzilli A, Pace A, Garramone F, Cavaliere C, Pardini M, Rizzetto C, Sorbi S, Perri R, Tiraboschi P, Canessa N, Cotelli M, Ferri R, Weintraub S, Marra C, Tagliavini F, Catricala E, Cappa SF. Italian adaptation of the Uniform Data Set Neuropsychological Test Battery (I-UDSNB 1.0): development and normative data. Alzheimers Res Ther. 2022 Aug 19;14(1):113. doi: 10.1186/s13195-022-01056-x. PMID 35982477
- [Background] Costa DSJ, Loh V, Birney DP, Dhillon HM, Fardell JE, Gessler D, Vardy JL. The Structure of the FACT-Cog v3 in Cancer Patients, Students, and Older Adults. J Pain Symptom Manage. 2018 Apr;55(4):1173-1178. doi: 10.1016/j.jpainsymman.2017.12.486. Epub 2017 Dec 30. PMID 29291932
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Fernandes HA, Richard NM, Edelstein K. Cognitive rehabilitation for cancer-related cognitive dysfunction: a systematic review. Support Care Cancer. 2019 Sep;27(9):3253-3279. doi: 10.1007/s00520-019-04866-2. Epub 2019 May 30. PMID 31147780
- [Background] Sullivan GM, Feinn R. Using Effect Size-or Why the P Value Is Not Enough. J Grad Med Educ. 2012 Sep;4(3):279-82. doi: 10.4300/JGME-D-12-00156.1. No abstract available. PMID 23997866
- [Background] Carey CL, Woods SP, Gonzalez R, Conover E, Marcotte TD, Grant I, Heaton RK; HNRC Group. Predictive validity of global deficit scores in detecting neuropsychological impairment in HIV infection. J Clin Exp Neuropsychol. 2004 May;26(3):307-19. doi: 10.1080/13803390490510031. PMID 15512922
- [Background] Costa A, Bagoj E, Monaco M, Zabberoni S, De Rosa S, Papantonio AM, Mundi C, Caltagirone C, Carlesimo GA. Standardization and normative data obtained in the Italian population for a new verbal fluency instrument, the phonemic/semantic alternate fluency test. Neurol Sci. 2014 Mar;35(3):365-72. doi: 10.1007/s10072-013-1520-8. Epub 2013 Aug 21. PMID 23963806
- [Background] Catricala E, Della Rosa PA, Ginex V, Mussetti Z, Plebani V, Cappa SF. An Italian battery for the assessment of semantic memory disorders. Neurol Sci. 2013 Jun;34(6):985-93. doi: 10.1007/s10072-012-1181-z. Epub 2012 Sep 9. PMID 22960873
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Caffarra P, Vezzadini G, Dieci F, Zonato F, Venneri A. Rey-Osterrieth complex figure: normative values in an Italian population sample. Neurol Sci. 2002 Mar;22(6):443-7. doi: 10.1007/s100720200003. PMID 11976975